CLINICAL TRIAL: NCT01595737
Title: Comparison of the Administration of Levosimendan and Placebo in the Preparation of Critical Patients for Heart Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ACA-SPAI-2008-20
Record Dates: First submitted 2012-05-07; First posted 2012-05-10 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2012-05

CONDITIONS: Cardiac Surgery
MeSH Terms: interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levosimendan (Experimental)
  Interventions: Drug: Levosimendan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levosimendan — Levosimendan perfusion for 12 hours before surgery by a single route, at a dosage of 0.1µg/kg/min without receiving the loading dose.
  Arms: Levosimendan
Drug: Placebo — Placebo group patients will receive a perfusion of 5% glucose solution. This clear solution, free of visible particles, will have 0.4mg of riboflavin sodium phosphate, 100mg of anhydrous alcohol and water for injection up to 1ml added to it. This solution will be calculated as a dose of 0.1µg/kg/min.
  Arms: Placebo

SUMMARY:
This study aims to examine the efficacy of levosimendan in terms of reducing postoperative mortality and severe morbidity in patients undergoing non-emergent surgery for coronary revascularisation with or without ischaemic mitral regurgitation and who may or may not require repair or replacement of the mitral valve and have a LVEF < 35%.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 years and < 85 years.
* LVEF ≤ 35%
* Indication for elective surgery for coronary revascularisation, with or without mitral valve repair.
* Freely choose to participate in trial and sign an informed consent

Exclusion Criteria:

* The patient does not accept the protocol.
* Allergy (hypersensitivity) to levosimendan, any of its components or to riboflavin.
* Severe hypotension or severe tachycardia prior to entering study.
* Significant mechanical obstruction affecting ventricular filling and/or emptying.
* History of Torsades.
* Requirement for inotropic or vasoactive drugs or any type of mechanical assistance for 48 hours prior to surgery.
* Onset of angina or acute myocardial infarction within 48 hours prior to surgery, or cardiogenic shock.
* Surgery needs that are different from those planned.
* Chronic or severe kidney failure requiring haemodialysis or peritoneal dialysis or creatinine clearance values below 30ml/min or presence of nephrotic syndrome.
* Liver failure with transaminases 4 times above the normal maximum value.
* The patient must undergo a concurrently scheduled surgery, such as for a valve other than the mitral.
* When a screening cannot be performed at least during the 24 hours before surgery.
* Uncontrolled diabetes mellitus (blood glucose > 24mmol/l or 432mg/dl).
* History of any disease over the last five years that may compromise the patient's life, other than their heart disease.
* The patient is currently abusing alcohol or toxic substances.
* Presence of any other medical or psychiatric condition that the researcher believes makes a candidate ineligible for the study.
* Women with childbearing potential who are not using an effective contraception method.
* Participation in the last 30 days in any other study with either experimental drugs or devices.
* Body Mass Index (BMI) greater than 35.
* Administration of levosimendan in the last 30 days.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days
  Rate of mortality
Morbidity | 30 days
  Rate of morbidity

SECONDARY OUTCOMES:
Dose of inotropic drugs used | 30 days
  Requirements for inotropic drugs
Dose of vasoactive drugs used | 30 days
  Requirements for vasoactive drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain